CLINICAL TRIAL: NCT06760689
Title: The Effect of Virtual Reality Glasses Used in Gynecologic Cancer Patients Receiving Chemotherapy on Treatment Compliance and Anxiety Level.
Brief Title: Brief Title- Virtual Reality Glasses in Gynecologic Cancer
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Beyza Önder, Nurse, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CAKU-HEM-BO-01
Record Dates: First submitted 2024-12-29; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Gynecologic Cancers; Anxiety
Keywords: Anxiety; chemotherapy; Gynecological cancer; Virtual reality; Adherence to treatment; rastgele kontrollü deneme
MeSH Terms: conditions — Anxiety Disorders; Treatment Adherence and Compliance | interventions — Weights and Measures

STUDY DESIGN:
Intervention Model Description: The study has a single-center, randomized controlled experimental design. It includes the experimental and control group.
Who Masked: Participant
Masking Description: It will be done bilaterally to determine whether there is a difference between the experimental and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The patient was given detailed information about the research and intervention, and written consent was obtained with an informed voluntary consent form. The patient's information was obtained through the descriptive information form containing sociodemographic information.The same ways were applied for 1,2,3 cures. The researcher applied the pre-test State and Trait Anxiety Scale, and the Chronic Disease Adaptation Scale (CHSS) to the patient.The patient was directed to move to the room designated by the nurse in the outpatient unit. Before the chemotherapy course began, the patient was shown the content that the patient could watch through virtual reality glasses on the phone.He was asked to choose one of them.The patient watched a video of his/her choice with the virtual reality glasses application (20 min). At the end, the glasses were removed. Afterwards, the State and Trait Anxiety Scale and the Chronic Diseases Adjustment Scale (CHAS) were applied.
  Interventions: Device: virtual reality glasses; Other: scale
- control group (Active Comparator): The pre-test State and Trait Anxiety Scale and Chronic Disease Adjustment Scale (CHAS) were applied to the patient by the researcher.
  The patient was directed to the room determined by the nurse in the outpatient treatment unit.
  The patient's chemotherapy infusion started.The patient received standard nursing care. After 30 minutes, the State and Trait Anxiety Scale and the Chronic Diseases Adjustment Scale (CHAS) were administered.
  Interventions: Other: scale

INTERVENTIONS:
Device: virtual reality glasses — One of the videos chosen by the patient will be opened in the virtual reality glasses and will be played for 20 minutes.
  Arms: Experimental group
Other: scale — The patient received standard nursing care. Scales were filled in after the course.

SUMMARY:
It was planned to determine the effect of virtual reality glasses used in female patients diagnosed with gynecological cancer and receiving chemotherapy on treatment compliance and anxiety level. The study has a single-center, randomized controlled experimental design.

DETAILED DESCRIPTION:
When cancer is diagnosed, a process of uncertainty begins for the individual. When an individual associates their illness with death, they often consider the situation to be frightening, painful, complex, and ambiguous, which can lead to mental confusion. ). In these emotional fluctuations, studies have revealed that a large proportion of patients experience various mental problems such as anxiety and anxiety disorders, coordination disorders and adherence to treatment, both due to the burden of the disease and the side effects of treatment. Emotional negativities felt by the patient may cause the recovery process to be prolonged, the quality of life to decrease, and the length of hospital stay to increase when in a hospital environment. In order to prevent such negativities, it is very important to identify the symptoms of anxiety and depression in cancer patients at an early stage and to initiate appropriate treatments. The development and application of the latest technology in the field of health offers new and non-invasive approaches to cancer-related symptom management. Virtual reality (SG), a new era in the management of symptoms, is the combination of fiction, imagination and reality, which is capable of real reflective animation at the same time under the control of many devices. Virtual reality (SG), a new era in the management of symptoms, is the combination of fiction, imagination and reality, which is capable of real reflective animation at the same time under the control of many devices.In a clinical study, it was concluded that distracting videos (tennis, boxing video, etc.) watched with virtual reality glasses had a beneficial therapeutic effect on edema.As a result of the one-week virtual reality application awareness training conducted on 50 women with ovarian cancer who experienced anxiety, depression and cancer-related fatigue during chemotherapy in Beijing, China, it was recorded that these symptoms improved significantly.When the literature was reviewed, it was predicted that the application of virtual reality glasses in cancer patients in our country was limited, and this study was planned to determine the effect of virtual reality glasses used in female patients diagnosed with gynecological cancer and receiving chemotherapy on the level of compliance and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old.
* Stage 1-2-3
* Knowing the disease diagnosis
* Knowing how to read and write in Turkish
* No history of seizures
* No cranial metastasis
* Not diagnosed with a psychiatric disorder, no dementia
* Those who receive their treatment in 21-day periods to ensure equality in application frequencies
* Able to use virtual reality glasses
* No visual or hearing impairment
* Volunteer patients

Exclusion Criteria:

* Stage 4
* Those with vertigo
* Those with hyperemesis during pregnancy
* Those who experience nausea and vomiting during travel
* Those with visual and hearing impairment
* Patients who do not know their cancer diagnosis, have been diagnosed with cancer but have not received treatment or have completed their cure

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals who have been diagnosed with gynecological cancer at the relevant institution, who will start their first course of chemotherapy, who have stage 1-2-3 cancer, who volunteer for the research, who are 18 years of age or older, and who are literate will be included.
Enrollment: 118 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Effect of Virtual Reality Glasses on Treatment Adherence and Anxiety Levels in Gynecological Cancer Patients Receiving Chemotherapy. | 20 weeks
  59 experimental groups of female patients in the outpatient chemotherapy unit will be shown a video of their choice, such as nature, underwater, or forest walk, placed in virtual reality glasses, taking into account the inclusion and exclusion criteria. Questions on two scales will be asked before and after this viewing. For the control group of 59 people, the same questions on two scales will be asked before and after chemotherapy without any intervention.
State and trait anxiety scale | 20 weeks
  This scale consists of two sub-dimensions, each consisting of 20 items, and contains a total of 40 items. The sub-scales are called "State Anxiety Scale" and "Trait Anxiety Scale". The first 20 items evaluate the emotional experiences of the individual in a certain situation. The emotions of the participants are expressed with the specific features of (1) None, (2) A Little, (3) A Lot, and (4) Completely. The items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20 in the State Anxiety Scale consist of translated expressions. These scores are translated in return (1=4, 2=3, 3=2, 4=1). Others represent correct objects. The state anxiety score varies between 20 and 80 in total, and reflects personal anxiety rates. High scores indicate high anxiety levels, and low scores indicate low anxiety levels.
Chronic Disease Adjustment Scale | 20 weeks
  It is a scale used to evaluate the adaptation level of patients with chronic diseases. This scale, which consists of three subdimensions and 25 items, measures physical adaptation with items 1, 9, 10, 13, 14, 15, 16, 18, 22, 23, and 24 (maximum 55, minimum 11 points), social adaptation with items 2, 3, 5, 7, 17, 19, and 25 (maximum 35, minimum 7 points) and psychological adaptation with items 4, 6, 8, 11, 12, 20, and 21 (maximum 35, minimum 7 points). The total score obtained from the scale is 125. High scores obtained from the subdimensions or the entire scale indicate that the patients' adaptation level to the disease is high.

CONTACTS AND LOCATIONS:
Locations (1):
- Etlik Şehir Hastanesi, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No